CLINICAL TRIAL: NCT07019649
Title: Tailoring Initial Type 2 Diabetes Care to Meet the Needs of Younger Latinx Adults: A Randomized Pilot Study
Brief Title: Randomized Pilot Trial of AYUDA Program for Younger Latinx Adults With Type 2 Diabetes
Acronym: AYUDA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2225114-1
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AYUDA Program (Experimental): Participants enrolled in the AYUDA program will receive text messages twice a week containing education and resources related to diabetes care and self-management, in addition to their usual diabetes care.
  Interventions: Behavioral: AYUDA Program
- Usual Care (No Intervention): No intervention will be employed. This arm will continue to receive their usual diabetes care.

INTERVENTIONS:
Behavioral: AYUDA Program — Participants randomized to the intervention arm will be enrolled in the AYUDA program, where they will receive text messages twice a week over 12 weeks containing diabetes education and self-management resources, including links to resources available to all KPNC members.
  Arms: AYUDA Program

SUMMARY:
The study will evaluate the feasibility, acceptability, and effectiveness of AYUDA (Assisting Younger Adults with Diabetes), a 12-week culturally text message program for Latinx adults newly diagnosed with type 2 diabetes who are caregivers to a child under 18 years old within Kaiser Permanente Northern California.

DETAILED DESCRIPTION:
After designing the AYUDA program with input from the people it is meant to help, we are conducting a randomized pilot study. This study will test the program with younger Latinx adults who have recently been diagnosed with type 2 diabetes and who are also caregivers for dependent children.

AYUDA is a health system specifically designed for this group, focusing on their life stage as young adults and their cultural background. The study will evaluate how well AYUDA helps participants reach important early blood sugar control goals, which can lead to better health over time and reduce complications.

ELIGIBILITY:
Inclusion Criteria:

* KPNC member, age >18 and age <45 with
* New clinical diagnosis of T2D within the prior 6 months
* Caregiver to at least one child <18 years of age at time of diabetes diagnosis
* Identifies at Latino/a/x
* Can receive text messages
* Proficient (written and spoken) in English or Spanish

Exclusion Criteria:

* Pregnant women
* Type 1 Diabetes

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-06-18 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Differences between study arms in HbA1c change 6-months following enrollment | 6-months following enrollment
  Change in HbA1c will be assessed using HbA1c values obtained through routine care, with the most recent HbA1c preceding study enrollment and the HbA1c value closest to 6-months following enrollment used to assess HbA1c change.

SECONDARY OUTCOMES:
Healthcare contact | 6-months following enrollment
  Differences in healthcare contact with members of the T2D diabetes care team, including care manager, PCPs, educators.
Completion of recommended HbA1c monitoring | 6-months following enrollment
  Completing HbA1c labs
T2D-related medication initiation | 6-months following enrollment
  Initiation of T2D-related medication
T2D-related medication adherence | 6-months following enrollment
  Adherence to T2D-related medication
Use of remote glucose monitoring to measure glucose levels | 6-months following enrollment
  Use of a remote glucose monitoring to measure glucose levels
Participant-reported measures: Diabetes distress | Study enrollment and 6-months following enrollment
  Assessed at study enrollment and 6-months following enrollment
Participant-reported measures: Motivation and locus of control | Study enrollment and 6-months following enrollment
  Assessed at study enrollment and 6-months following enrollment
Participant-reported measures: Care Experience | Study enrollment and 6-months following enrollment
  Assessed at study enrollment and 6-months following enrollment
Participant-reported measures: Children's Behaviors | Study enrollment and 6-months following enrollment
  Assessed at study enrollment and 6-months following enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Northern California, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No